CLINICAL TRIAL: NCT06662006
Title: Efficacy and Safety of Second-line Therapy by Nal-IRI/5-FU/LV Chemotherapy Combined With PD-L1 Inhibitor and Multi-target Anti-angiogenic Small Molecule±SBRT in Metastatic Pancreatic Cancer Patients: a Prospective, Multicentre, Single-arm, Multi-cohort Study
Brief Title: Nal-IRI/5-FU/LV Chemotherapy Combined With PD-L1 Inhibitor and Multi-target Anti-angiogenic Small Molecule±SBRT as Second-line Therapy in Metastatic Pancreatic Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-OBU-JS-PanC-II-015
Record Dates: First submitted 2024-10-17; First posted 2024-10-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Advanced Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; liposomal irinotecan; benmelstobart; anlotinib
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nal-IRI/5-FU/LV + benmelstobart + anlotinib ± SBRT (Experimental): liposomal irinotecan (nal-IRI) plus 5-fluorouracil (5-FU)/leucovorin (LV) (nal-IRI/5-FU/LV) combined with benmelstobart and anlotinib ± SBRT
  Interventions: Drug: nal-IRI,5-fu,LV, benmelstobart, anlotinib

INTERVENTIONS:
Drug: nal-IRI,5-fu,LV, benmelstobart, anlotinib — liposomal irinotecan (nal-IRI) plus 5-fluorouracil (5-FU)/leucovorin (LV) (nal-IRI/5-FU/LV) combined with benmelstobart and anlotinib ± SBRT

SUMMARY:
This study is a single-arm, multi-center, multi-cohort, prospective clinical study initiated by the investigator.

The indication of this study is: patients with advanced metastatic pancreatic cancer who have progressed after first-line chemotherapy. Eligible patients will be assigned to liposomal irinotecan (nal-IRI) plus 5-fluorouracil (5-FU)/leucovorin (LV) (nal-IRI/5-FU/LV) combined with benmelstobart and anlotinib ± SBRT.

The total sample size for this study is expected to be 56 subjects.

DETAILED DESCRIPTION:
For patients with advanced metastatic pancreatic cancer who failed first-line treatment, the screening and enrollment will be completed according to the enrollment and exclusion criteria described in the study protocol, and the informed consent form will be signed after full communication. After enrollment, patients will be treated with cohort A) or cohort B), and followed up regularly.

Cohort A: nal-IRI/5-FU/LV + PD-L1 inhibitor + multi-target anti-angiogenic small molecule:

Irinotecan liposome: 50mg/m2 IV D1, D15 LV: 400mg/m2 IV D1, D15 5-FU ：2.4g/m2 CIV 46h D1, D15 bemosubaemab: 1200mg IV Q3W Anlotinib: 12mg po D1-D14 Q3W

Cohort B: nal-IRI/5-FU/LV + PD-L1 inhibitor+ multi-target anti-angiogenic small molecule+SBRT Group:

Irinotecan liposomes: 50mg/m2 IV D1, D15 LV: 400mg/m2 IV D1, D15 5-FU ：2.4g/m2 CIV 46h D1, D15 bemosubaemab: 1200mg IV Q3W Anlotinib: 12mg po D1-D14 Q3W SBRT

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years, ECOG score of ≤2 points, expected survival time ≥ 3 months.
2. Patients with histologically or cytologically confirmed advanced metastatic pancreatic cancer.
3. Imaging suggests distant measurable lesions.
4. Failure of first-line therapy and no use of fluorouracil, irinotecan, or liposomal irinotecan drugs in the first-line therapy.

Patients need to meet the following hematologic indicators e1. Neutrophil count ≥ 1.5×109/L e2. Hemoglobin ≥ 10 g/dL e3. Platelet count ≥ 100×109/L f. Patients need to meet the following biochemical parameters f1. Total bilirubin ≤ 1.5× upper limit of normal (ULN) f2. AST and ALT <1.5×ULN f3. Creatinine clearance ≥ 60ml/min g. Patients of childbearing age need to take appropriate protective measures (contraception or other methods of birth control) before enrollment and during the trial.

H. Has signed an informed consent form. i. Able to follow the study protocol and follow-up process.

Exclusion Criteria:

1. Have received second-line or more anti-tumor therapy in the past.
2. First-line treatment with fluorouracil, irinotecan or liposomal irinotecan, etc.
3. Patient has a prior history of other tumors, unless it is cervical cancer in situ, treated squamous cell carcinoma or bladder epithelial tumors (Ta and TIS) or other malignancies that have received curative therapy (at least more than 5 years prior to enrollment).
4. Patient has an active bacterial or fungal infection (≥ 3rd edition NCI-CTC2 grade).

Patient has HIV, HCV, HBV infection, uncontrolled coronary artery disease or asthma, uncontrolled cerebrovascular disease or other disease deemed non-enrollable by the investigator.

f. Patients with autoimmune diseases or immunodeficiencies who should be treated with immunosuppressive drugs.

g. Pregnant and lactating women. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.

h. Substance abuse, clinical or psychological, or social factors that compromise informed consent or study conduct.

i. Those who may be allergic to treatment drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective effective rate (ORR) | 28 days per cycle, with ≤6 cycles of treatment expected per patient
  The overall response rate, including complete response (CR) + partial response (PR), refers to the proportion of patients whose tumor shrinks to a certain amount and remains for a certain period of time.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 28 days per cycle, with ≤6 cycles of treatment expected per patient
  Refers to the proportion of patients whose tumors have shrunk or stable and remain for a certain period of time, including complete remission (CR), partial remission (PR) and stable (SD) cases.
Median overall survival (mOS) | 28 days per cycle, with ≤6 cycles of treatment expected per patient
  Refers to the numerical value in which the survival time of all patients is arranged in the order from smallest to largest in clinical research, and is located in the middle position.
Median progression-free survival (mPFS) | 28 days per cycle, with ≤6 cycles of treatment expected per patient
  Refers to the value in which all patients are sorted according to the length of progression-free survival time in clinical studies, and is located in the middle position.

OTHER OUTCOMES:
Exploring potential efficacy prediction biomarkers | 28 days per cycle, with ≤6 cycles of treatment expected per patient
  Explore potential efficacy prediction biomarkers: including patients' tumor-related serological indicators, such as peripheral blood lymphocyte count, twelve cytokine tests (IL-2, IFN-γ, TNF-α, IL-4, IL-5, IL6, IL-10, IL-17, IL-1β, IL-8, IFN-α, IL-12p70) and ctDNA detection. This type of index was collected once at the baseline of the patient, and again after every 2 cycles of treatment until the patient entered the maintenance phase or the disease progressed.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No